CLINICAL TRIAL: NCT03349177
Title: Pathological Complete Response Rate in Locally Advanced Breast Cancer With Neoadjuvant Fluorourcil/Epirubicin/Cyclophosphamide, Epirubicin/Cyclophosphamide Followed by Docetaxel, or Docetaxel/Cyclophosphamide as Neoadjuvant Chemotherapy
Brief Title: Pathological Complete Response Rate in Locally Advanced Breast Cancer With FEC, EC-T, or TC as Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhiyong Yu (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Yu, Director of the Breast Surgery Ⅰ, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI-02
Record Dates: First submitted 2017-10-14; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Pathological Complete Response; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Doxorubicin; Fluorouracil; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- FEC group (Experimental): Fluorouracil 500mg/m2 on day 1, epirubicin 100mg/m2 on day 1 and cyclophosphamide 500mg/m2 on day 1 every 3 weeks for six cycles
  Interventions: Drug: Epirubicin; Drug: Fluorouracil; Drug: Cyclophosphamide
- EC-T group (Experimental): Epirubicin 100mg/m2 on day 1 cyclophosphamide 600mg/m2 on day1 every 2 weeks for four cycles followed by docetaxel 100mg/m2 on day 1 every 3 weeks for four cycles
  Interventions: Drug: Epirubicin; Drug: Docetaxel; Drug: Cyclophosphamide
- TC group (Experimental): Docetaxel 75mg/m2 on day 1 and cyclophosphamide 600mg/m2 on day 1 every 3 weeks for six cycles
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Epirubicin — 100mg/m2
  Other Names: Adriacin
  Arms: EC-T group; FEC group
Drug: Fluorouracil — 500mg/m2
  Other Names: Fluorouracil injection
  Arms: FEC group
Drug: Docetaxel — 75mg/m2(TC), 100mg/m2(EC-T)
  Other Names: Docetaxel injection
  Arms: EC-T group; TC group
Drug: Cyclophosphamide — 500mg/m2(FEC), 600mg/m2(EC-T and TC)
  Other Names: Cyclophosphamide injection

SUMMARY:
Neoadjuvant chemotherapy (NAC) has become the standard therapy for both locally advanced and early-stage breast cancer in recent years for the improvement breast conserving surgery rate and the evaluation of treatment response in vivo. Pathological complete response (pCR) is an independent prognostic factor irrespective of breast cancer intrinsic subtypes after NAC. The trial is designed to compare effectiveness between anthracycline and/or taxane as neoadjuvant chemotherapy for operable advanced breast cancer in different molecular typing. In this trial the investigators will randomly assign 200 primary breast cancer patients to receive six cycles of fluorourcil, epirubicin,and cyclophosphamide(FEC), or four cycles of epirubicin and cyclophosphamide (EC) followed by four cycles of docetaxel(T), or six cycles of docetaxel and cyclophosphamide (TC). Trasuzumab was recommended combining docetaxel to patients if HER-2 positive.The effectiveness of therapy will be estimated after every two cycles of neoadjuvant chemotherapy. Surgery will be performed after completing designated full cycles of neoadjuvant chemotherapy. The primary endpoint is to assess pathologic complete response (pCR, ypT0/is ypN0) rate in different regiments. The secondary endpoint is to assess the relationship between pCR rate with molecular typing in different regiments, so that the investigators could optimize neoadjuvant chemotherapy regiment according to molecular typing.

DETAILED DESCRIPTION:
The trial is designed to compare effectiveness between anthracycline and/or taxane as neoadjuvant chemotherapy for operable advanced breast cancer in different molecular typing. In this trial the investigators will randomly assign 200 primary breast cancer patients to receive six cycles of fluorourcil, epirubicin,and cyclophosphamide(FEC), or four cycles of epirubicin and cyclophosphamide (EC) followed by four cycles of docetaxel(T), or six cycles of docetaxel and cyclophosphamide (TC). Trasuzumab was recommended combining docetaxel to patients if HER-2 positive.The effectiveness of therapy will be estimated after every two cycles of neoadjuvant chemotherapy. Surgery will be performed after completing designated full cycles of neoadjuvant chemotherapy. The primary endpoint is to assess pathologic complete response (pCR, ypT0/is ypN0) rate in different regiments. The secondary endpoint is to assess the relationship between pCR rate with molecular typing in different regiments, so that the investigators could optimize neoadjuvant chemotherapy regiment according to molecular typing.

ELIGIBILITY:
Inclusion Criteria:

* All patients were required to give written informed consent.
* Patients present with operable breast cancers that were diagnosed by histopathology and have no distant metastasis.
* Have no history of anti-cancer therapies including chemotherapy, radiation therapy, hormone therapy and surgical therapy.
* Have normal cardiac functions by echocardiography.
* ECOG scores are ≤ 0-1.
* Patients are disposed to practice contraception during the whole trial.
* The results of patients' blood tests are as follows:

Hb ≥ 90 g/L WBC ≥ 3.0×109/L Plt ≥ 100×109/L Neutrophils ≥ 1.5×109/L ALT and AST ≤ 2.5 times of normal upper limit. TBIL ≤ 1.5 times of normal upper limit. Creatinine ≤ 1.5 times of normal upper limit.

Exclusion Criteria:

* Have other cancers at the same time or have the history of other cancers in recent five years, excluding the controlled skin basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of cervix.
* Active infections
* Severe non-cancerous diseases.
* The patients are undergoing current administration of anti-cancer therapies, or are attending some other clinical trails.
* Inflammatory breast cancer.
* Pregnant or lactational, or patients refuse to practice contraception during the whole trial.
* The patients are in some special conditions that they can't understand the written informed consent, such as they are demented or hawkish.
* Have allergic history of the chemotherapeutic agents.
* Bilateral breast cancers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2017-11-27 (Estimated); Primary Completion 2019-11-27 (Estimated); Study Completion 2019-11-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Pathological Complete Response (pCR) | 2 years
  Participants were evaluated following eight cycles of treatment and after surgery to assess for pCR. pCR was defined as no invasive or in situ residual tumor masses in the breast and lymph nodes according to pathologist examination. The percentage of participants with pCR was reported, and the 95% CI for one-sample binomial was constructed using the Pearson-Clopper method.

SECONDARY OUTCOMES:
The relation between pCR rate, molecular subtypes, and different regiments. | 2 years
  The correlations were calculated using the Spearman rank correlation coefficient. The criteria for judging the size of the correlation coefficient were applied: correlations<0.30 are considered minor, correlations between 0.3-0.49 are considered medium, and ≥0.5 are considered strong. Cohen's kappa statistic was used to determine inter-examiner agreement. According to Altman's guidelines, it is poor when kappa scores ≤0.20, fair when kappa between 0.21-0.40, moderate when kappa between 0.41-0.60, good when kappa 0.61-0.80, and very good when kappa ≥0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Yu, PhD, Study Chair — Shandong Cancer Hospital and Institute; Xiaoshan Cao, MD, Principal Investigator — Shandong Cancer Hospital and Institute